CLINICAL TRIAL: NCT06799481
Title: Virtually Delivered Home-Based Exercise Intervention on Cognitive Impairment and Gut Microbiome in Adolescent and Young Adult Brain Tumor Survivors: A Pilot Randomized Controlled Trial
Brief Title: Virtual Home-based Exercise Intervention (RISE) to Improve Cancer-Related Cognitive Impairment and Gut Microbiome in Adolescent and Young Adult Brain Tumor Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Principal Investigator, Jinbing Bai, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00008229; NCI-2025-00181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008229 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6364-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer-related Cognitive Dysfunction; Primary Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Exercise; Behavior Therapy; Chromatin Immunoprecipitation Sequencing; Follow-Up Studies; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: To maintain blinding, only the exercise trainer and statistician will know group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (RISE) (Experimental): Patients receive access to Physitrack and participate in personalized, progressive aerobic training over 30-40 minutes 3-5 days a week and strength training exercises 2 days a week for 12 weeks. Patients also receive active lifestyle behavior coaching over 10 minutes on 2 days a week for weeks 1-4 and then once weekly for weeks 5-12.
  Interventions: Other: Aerobic Exercise; Behavioral: Behavioral Intervention; Other: Internet-Based Intervention; Other: Questionnaire Administration; Other: Resistance Training
- Arm II (attention control) (Active Comparator): Patients receive calls from the trainer once weekly for 12 weeks. Patients also wear a Fitbit for 7 days at baseline to week 12.
  Interventions: Procedure: Follow-Up; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Aerobic Exercise — Participate in personalized, progressive aerobic training
  Other Names: Aerobic Activity
  Arms: Arm I (RISE)
Behavioral: Behavioral Intervention — Receive active lifestyle behavior coaching
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (RISE)
Procedure: Follow-Up — Receive calls from the trainer
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
  Arms: Arm II (attention control)
Other: Internet-Based Intervention — Receive access to Physitrack
  Arms: Arm I (RISE)
Other: Medical Device Usage and Evaluation — Wear a Fitbit monitor
  Arms: Arm II (attention control)
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Participating in strength training exercises
  Other Names: Strength Training
  Arms: Arm I (RISE)

SUMMARY:
This clinical trial evaluates the impact of a research intervention of virtually supervised exercise program (RISE) on cancer-related cognitive impairment (CRCI), physical activity in adolescent and young adult (AYA) brain tumor survivors. This clinical trial also evaluates the impact of RISE on the collection of microorganisms that exist in the intestines (gut microbiome). Up to 45% of AYA brain tumor survivors experience CRCI, including issues with attention and memory. CRCI can have a negative impact on education, independent living and can worsen long-term quality of life. Moderate-intensity levels of exercise, particularly aerobic and resistance training, have been shown to improve cognitive function. Additionally, exercise can change the composition and function of the gut microbiome, which may lead to improved cognitive function. Unfortunately, only about 50% of AYAs with cancer receive exercise information or meet the physical activity recommendations. Tailoring a virtually delivered exercise intervention to meet the unique needs of AYAs may improve access to exercise. Participating in the virtual home-based exercise intervention, RISE, may improve physical activity and cognitive impairment in AYA brain tumor survivors and may also help researchers understand the relationship of exercise on the gut microbiome and cognitive function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of conducting a two-site pilot randomized controlled trial (RCT) to test the RISE in AYA brain tumor survivors.

II. Examine the impact of RISE on CRCI (primary) and physical activity (secondary).

EXPLORATORY OBJECTIVE:

I. Explore the impact of RISE on the gut microbiome diversity and composition.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (RISE INTERVENTION): Patients receive access to Physitrack and participate in personalized, progressive aerobic training over 30-40 minutes 3-5 days a week and strength training exercises 2 days a week for 12 weeks. Patients also receive active lifestyle behavior coaching over 10 minutes on 2 days a week for weeks 1-4 and then once weekly for weeks 5-12.

ARM II (ATTENTION CONTROL): Patients receive calls from the trainer once weekly for 12 weeks. Patients also wear a Fitbit for 7 days at baseline to week 12.

After completion of study intervention, patients are followed up at week 18.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-39 years
* With primary brain tumor with cranial radiotherapy
* 6 months to 4 years post cranial radiotherapy
* Functional Assessment of Cancer Therapy (FACT)-Cognitive Function score < 60 based on self-report (used among AYAs with non-neural cancer)
* Able to provide informed consent/assent
* Able to walk and receive clearance from a provider to participate based on the Physical Activity Readiness Questionnaire
* Currently engaging in < 150 minutes of physical activity per week
* Willing to use smartphone-based applications (app)

Exclusion Criteria:

* Secondary malignancies, germline genetic syndrome, or recurrent disease requiring re-irradiation of the brain
* Moderate to severe traumatic brain injury with brain damage beyond that expected from brain tumor and treatment
* Developmental disorders (e.g., autism) or major psychotic illness (e.g., schizophrenia, depression) to avoid confounding impact related to these disorders

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Up to 1.5 years
  Feasibility will be ≥ 50% enrollment of eligible survivors. Descriptive statistics (e.g., frequency and percentage) will be used.
Adherence to research intervention of virtually supervised exercise program (RISE) | Up to 12 weeks
  Feasibility will be ≥ 75% adherence to RISE. Descriptive statistics (e.g., frequency and percentage) will be used.
Retention | Up to 12 weeks
  Feasibility will be ≥ 80% retention at end of intervention. Descriptive statistics (e.g., frequency and percentage) will be used.
Acceptability | Up to 18 weeks
  Will use an 11-item acceptability questionnaire. A ≥ 4 ("agree" to "strongly agree") per item equates to acceptability. Descriptive statistics (e.g., frequency and percentage) will be used.
Change in physical activity levels | Baseline up to 18 weeks
  Will be measured by Fitbit. Physical activity estimates considered as valid if the monitor is worn ≥ 10 hours/day on ≥ 4 days. Will use mixed-effect analysis of variance to model the correlation with timepoint and treatment group plus interaction if applicable, clustering on patient to control for repeated measures, and controlling for baseline measure and other covariates, which are considered prognostic or differ at baseline. A 95% level of statistical confidence will be assumed in all statistical testing.
Change in cancer-related cognitive impairment | Baseline up to 18 weeks
  Will use mixed-effect analysis of variance to model the correlation with timepoint and treatment group plus interaction if applicable, clustering on patient to control for repeated measures, and controlling for baseline measure and other covariates, which are considered prognostic or differ at baseline. A 95% level of statistical confidence will be assumed in all statistical testing.

SECONDARY OUTCOMES:
Gut microbiome | Up to 18 weeks
  Fecal specimens will be collected for the gut microbiome. Will use mixed-effect analysis of variance to model the correlation with timepoint and treatment group plus interaction if applicable, clustering on patient to control for repeated measures, and controlling for baseline measure and other covariates, which are considered prognostic or differ at baseline. A 95% level of statistical confidence will be assumed in all statistical testing.
Physical function | At baseline and at 12 and 18 weeks
  Will use mixed-effect analysis of variance to model the correlation with timepoint and treatment group plus interaction if applicable, clustering on patient to control for repeated measures, and controlling for baseline measure and other covariates, which are considered prognostic or differ at baseline. A 95% level of statistical confidence will be assumed in all statistical testing.
Patient Quality of Life | At baseline and at 12 and 18 weeks
  Will be assessed by Patient Reported Outcomes Measurement Information System-29 recommended. Will use mixed-effect analysis of variance to model the correlation with timepoint and treatment group plus interaction if applicable, clustering on patient to control for repeated measures, and controlling for baseline measure and other covariates, which are considered prognostic or differ at baseline. A 95% level of statistical confidence will be assumed in all statistical testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbing Bai, PhD, RN, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - MD Anderson Cancer Center, Houston, Texas